CLINICAL TRIAL: NCT02395978
Title: A Phase II Study of PDC-1421 Capsule to Evaluate the Safety and Efficacy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Phase II BLI-1005-002
Record Dates: First submitted 2014-09-17; First posted 2015-03-24 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2019-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Part I is a open label, dose escalation with two dosage levels study. Part II is a randomized (1:1:1), double-blind, placebo-controlled, parallel groups with three treatment arms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part I: 1 PDC-1421 Capsule (Experimental): 1 PDC-1421 Capsule TID, p.o. after meal for 28 days
  Interventions: Drug: PDC-1421 Capsule
- Part I: 2 PDC-1421 Capsule (Experimental): 2 PDC-1421 Capsule TID, p.o. after meal for 28 days
  Interventions: Drug: PDC-1421 Capsule
- Part II: 2 PDC-1421 Capsule (Experimental): 2 PDC-1421 Capsule TID, p.o. after meal for 42 days
  Interventions: Drug: PDC-1421 Capsule
- Part II: 1 PDC-1421 Capsule plus 1 placebo (Experimental): 1 PDC-1421 Capsule plus 1 placebo TID, p.o. after meal for 42 days
  Interventions: Drug: PDC-1421 Capsule; Drug: placebo
- Part II: 2 placebo (Placebo Comparator): 2 placebo TID, p.o. after meal for 42 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PDC-1421 Capsule — PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.
  Other Names: BLI-1005
  Arms: Part I: 1 PDC-1421 Capsule; Part I: 2 PDC-1421 Capsule; Part II: 1 PDC-1421 Capsule plus 1 placebo; Part II: 2 PDC-1421 Capsule
Drug: placebo — Placebo contained corn starch.
  Arms: Part II: 1 PDC-1421 Capsule plus 1 placebo; Part II: 2 placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy in patients with major depressive disorder.

DETAILED DESCRIPTION:
The screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The following study will be conducted in two parts. Part I is an open-label study, multiple center and dose escalation evaluation in twelve patients. Six subjects each will be evaluated for safety and efficacy assessments at 1 or 2 capsules TID dose for 28 days, sequentially. Each of them will be assessed twice in the first week after administration of PDC-1421 Capsules and once a week in the following treatment.

Part II is a randomized, double-blind, placebo-controlled, parallel-group study. 60 subjects will be randomly assigned on a 1:1:1 basis to one of the three arms (1 PDC-1421 Capsule plus 1 placebo TID, 2 PDC-1421 Capsules TID, 2 placebo TID) for 6 weeks and evaluated the safety and efficacy every two weeks during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients aged 20-65 years
2. Subjects must be able to understand and willing to sign informed consent
3. Female subjects of child-bearing potential must test negative to pregnancy and use appropriate birth control method from the beginning of study to the 15 days later after ending of study
4. Met criteria for MDD without psychotic features as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision® (DSM-IV-TR) and confirmed by use of the Mini International Neuropsychiatric Interview (MINI).
5. 17-item HAM-D (Hamilton Rating Scale for Depression) total score ≧20 and CGI (Clinical Global Impression) total score ≧4

Exclusion Criteria:

1. Have a current or previous major psychiatric disorders which be defined to be per the DSM-IV-TR, including obsessive-compulsive disorder, posttraumatic stress disorder, bipolar I or II, manic or hypomanic episode, schizophrenia, major Axis II disorders which might compromise the study, and major depression with psychotic symptoms, mental retardation.
2. Use of any treatment for MDD in the last 2 weeks before visit 1 (4 weeks for fluoxetine).
3. Use of psychoactive drugs within the last 2 weeks before visit 1 other than that subjects had insomnia who need the treatment as determined by the Investigator.
4. Subjects who were non-responsive to two or more courses of antidepressant medications given an adequate dosage for symptom treatment within four weeks, or by the judgment of the investigator considered to have treatment resistant depression (TRD), or a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS) or psychosurgery within the last year.
5. Have a history of any seizure disorder.
6. Any clinically significant abnormal vital sign, ECG, laboratory values as determined by the investigator which might interfere with the study.
7. Any organic disorder caused u medical related depression which cannot be under well-controlled such as clinically significant in neurological, gastrointestinal, renal, hepatic, cardiovascular, respiratory, metabolic, endocrine, hematological or other major disorders
8. Have a high suicidal risk as measured by MINI.
9. Have a history of substance abuse within the past 6 months or a positive urine drug screen for any substance of abuse at visit 1.
10. Have a history of severe allergies to more than 1 class of medication or multiple adverse drug reactions.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard King, Ph.D., Study Director — American BriVision Corporation
Locations (5):
- Stanford Depression Research Clinic, San Francisco, California, United States
- Taiwan (4):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Neihu Main Facility, Taipei
  - Wan Fang Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were recruited over a 49-month period from April of 2015 to March of 2019 at 5 studies sites in Taiwan and 1 study site in the United States.
Groups:
- Part I: 1 PDC-1421 Capsule: 1 PDC-1421 Capsule thrice daily (TID), oral administration (p.o.) after meal for 28 days
- Part II: 2 PDC-1421 Capsule: 2 PDC-1421 Capsule TID, p.o. after meal for 42 days
  PDC-1421 Capsule
- Part II: 1 PDC-1421 Capsule Plus 1 Placebo: 1 PDC-1421 Capsule plus 1 placebo TID, p.o. after meal for 42 days
  PDC-1421 Capsule
  placebo
- Part II: 2 Placebo: 2 placebo TID, p.o. after meal for 42 days
  placebo
Period: Overall Study
Arm/Group | Part I: 1 PDC-1421 Capsule | Part I: 2 PDC-1421 Capsule | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Started | 6 | 6 | 21 | 19 | 20
Completed | 6 | 6 | 19 | 14 | 15
Not Completed | 0 | 0 | 2 | 5 | 5

BASELINE CHARACTERISTICS:
Population: The ITT population included 12 subjects in Part I and 60 subjects in Part II. The PP population included 11 subjects in Part I and 44 subjects in Part II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I: 1 PDC-1421 Capsule | Part I: 2 PDC-1421 Capsule | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo | Total
Number analyzed (Participants) | 6 | 6 | 21 | 19 | 20 | 72
Age, Continuous [Mean (Full Range); unit: years] | 38.7 [20 to 48] | 43.2 [20 to 61] | 43.1 [20 to 64] | 42.1 [21 to 64] | 43.9 [20 to 64] | 42.7 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 8 | 6 | 8 | 27
  Male | 3 | 4 | 13 | 13 | 12 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 3 | 3 | 4 | 10
  Taiwan | 6 | 6 | 18 | 16 | 16 | 62
Weight [Mean (Full Range); unit: Kg] | 60.3 [45 to 74] | 61.1 [45.7 to 89] | 63 [35 to 103.9] | 59.2 [39.6 to 78.3] | 65 [45.3 to 103.4] | 62.2 [35 to 103.9]
Height [Mean (Full Range); unit: cm] | 162.5 [152 to 175] | 164.05 [151.4 to 178] | 163.8 [153 to 180] | 162.5 [144.8 to 184.2] | 165.2 [148 to 178] | 163.7 [144.8 to 184.2]

OUTCOME MEASURES:

1. Primary Outcome: Change of Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Week 6 Compared to Placebo for Part II.
Description: The MADRS is a 10-item checklist of depressive symptoms. Each Item is rated on a scale of 0-6, with anchors at 2-point intervals; higher scores indicating more severity (i.e., ranging from 0 [no sadness] to 6 extremely despondent]). The total MADRS score was calculated by summing the ratings of all items. The total MADRS score for this measure ranges from 0 (absence of symptoms) to 60 (maximum severity).
Time Frame: From Baseline to Week 6
Population: The Intention-To-Treat (ITT) population consisted of 60 randomized subjects. The Per-Protocol (PP) population consisted of 44 randomized subjects. This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  ITT population | -13.19 (9.68) | -9.21 (8.32) | -9.2 (7.98)
  PP population: number analyzed (Participants) | 15 | 15 | 14
  PP population | -13.4 (9.7) | -10.4 (5.18) | -8.6 (7.61)
Statistical Analysis 1: Comparison: Part II: 2 PDC-1421 Capsule vs Part II: 1 PDC-1421 Capsule Plus 1 Placebo vs Part II: 2 Placebo; Test type: Superiority; p = 0.393, Kruskal-Wallis

2. Secondary Outcome: Change of Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Week 2, 4 and 7 Part II.
Description: as for outcome 1
Time Frame: From Baseline to Week 2, 4, 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  From baseline to Week 2 | -7.4 (5.08) | -6.4 (8.87) | -5.5 (5.76)
  From baseline to Week 4 | -10.8 (7.95) | -7.6 (9.12) | -8.7 (7.07)
  From baseline to Week 7 | -13.6 (8.98) | -8.2 (7.99) | -9.9 (7.32)

3. Secondary Outcome: Change of Hamilton Depression Rating Scale (HAM-D-17) Total Score From Baseline to Week 2, 4, 6 and 7 for Part II.
Description: HAM-D-17 scale is a clinician rated scale comprised of 17 items aimed at assessing depression severity among patients for treatment. Each item on the questionnaire is scored on a 3 point (8 items) or 5 point (9 items) scale, depending on the item. The total HAM-D-17 score was calculated by summing the ratings of all items. . The highest possible score was 52, which represented the most severe measure of depression; the lowest possible score was 0, which represented an absence of depression.
Time Frame: From Baseline to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  From baseline to Week 2 | -7.9 (4.72) | -6.5 (6.22) | -4.3 (4.58)
  From baseline to Week 4 | -9.7 (6.03) | -7.5 (6.64) | -8.2 (4.72)
  From baseline to Week 6 | -11.0 (6.71) | -8.8 (7.21) | -8.7 (6.91)
  From baseline to Week 7 | -10.4 (6.23) | -7.9 (7.05) | -8.7 (5.95)

4. Secondary Outcome: Change of Hamilton Anxiety Rating Scale (HAM-A) Total Score From Baseline to Week 2, 4, 6 and 7 for Part II.
Description: HAM-A is a series of questions related to symptoms of anxiety. It rates the individual on a five-point scale (0~4) for each of the 14 items. Seven of the items specifically address psychic anxiety and the remaining seven items address somatic anxiety. The total HAM-A score was calculated by summing the ratings of all items. The total HAM-A score ranges from 0 to 56. The higher score represented a more severe measure of anxiety.
Time Frame: From Baseline to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  From baseline to Week 2 | -5.4 (3.06) | -4.3 (5.45) | -2.9 (4.66)
  From baseline to Week 4 | -7.2 (5.95) | -5.5 (6.55) | -6.2 (4.82)
  From baseline to Week 6 | -8.7 (6.04) | -7.0 (7.46) | -6.2 (6.30)
  From baseline to Week 7 | -8.9 (5.82) | -5.1 (7.15) | -6.6 (6.15)

5. Secondary Outcome: Change of Depression and Somatic Symptoms Scale (DSSS) From Baseline to Week 2, 4, 6 and 7 for Part II
Description: DSSS includes a simultaneous measure of depression and somatic symptoms that two issues frequently co-occur. Consisting of 22 items, the DSSS includes 12 depression-related items (even items + item-21) and 10 somatic items (add items without item-21) - 5 of which query pain symptoms(item-1, 7, 11, 13, 17), forming a pain sub-scale. Each Item is rated on a scale of 0 (Absent) - 3 (Severe).
  DSSS Depression Sub-Score was calculated by summing the 12 depression-related items with ranges from 0 (absence of symptoms) to 36 (maximum severity).
  DSSS Somatic Sub-Score was calculated by summing the 10 somatin-related items with ranges from 0 (absence of symptoms) to 30 (maximum severity).
  DSSS Pain Sub-Score was calculated by summing the 5 pain-related items with ranges from 0 (absence of symptoms) to 15 (maximum severity).
Time Frame: From Baseline to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  DSSS Depression Sub-Score- From baseline to Week 2 | -3.6 (5.26) | -3.1 (6.35) | -1.7 (3.15)
  DSSS Depression Sub-Score- From baseline to Week 4 | -4.5 (5.36) | -5.6 (5.58) | -4.0 (5.20)
  DSSS Depression Sub-Score- From baseline to Week 6 | -4.7 (7.71) | -5.9 (5.18) | -3.6 (5.09)
  DSSS Depression Sub-Score- From baseline to Week 7 | -5.4 (6.46) | -5.4 (5.46) | -3.3 (5.51)
  DSSS Somatic Sub-Score- From baseline to Week 2 | -2.3 (4.56) | -2.2 (4.11) | -1.1 (2.74)
  DSSS Somatic Sub-Score- From baseline to Week 4 | -2.6 (5.3) | -3.3 (3.38) | -0.9 (2.21)
  DSSS Somatic Sub-Score- From baseline to Week 6 | -2.9 (6.24) | -3.3 (3.94) | -2.3 (2.31)
  DSSS Somatic Sub-Score- From baseline to Week 7 | -3.1 (4.90) | -3.2 (2.94) | -1.3 (2.62)
  DSSS Pain Sub-Score- From baseline to Week 2 | -0.9 (2.46) | -1.0 (2.36) | -0.4 (2.01)
  DSSS Pain Sub-Score- From baseline to Week 4 | -1.2 (2.79) | -1.4 (2.01) | -0.6 (1.93)
  DSSS Pain Sub-Score- From baseline to Week 6 | -1.3 (3.23) | -1.4 (1.89) | -1.2 (1.76)
  DSSS Pain Sub-Score- From baseline to Week 7 | -1.3 (2.41) | -1.3 (1.60) | -0.5 (1.88)

6. Secondary Outcome: Change of Clinical Global Impression Scale - Severity (CGI-S) From Baseline to Week 2, 4, 6 and 7 for Part II.
Description: CGI-Severity (CGI-S) is a 7-point scale which rates illness severity of psychopathology from 1 (normal, not at all ill) to 7 (among the most extremely ill).
Time Frame: From Baseline to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  From baseline to Week 2 | -0.6 (0.50) | -0.7 (0.95) | -0.3 (0.57)
  From baseline to Week 4 | -1.1 (0.77) | -0.9 (1.2) | -0.9 (0.72)
  From baseline to Week 6 | -1.3 (1.20) | -1.0 (1.00) | -0.9 (1.02)
  From baseline to Week 7 | -1.4 (1.12) | -1.1 (0.99) | -1.0 (0.89)

7. Secondary Outcome: Percentage of Responders and Partial Responders in MADRS by Week 2, 4, 6 and 7 Weeks for Part II.
Description: Responder defined as a participant with ≧50% decrease from baseline in total score.
  Partial responder defined as a participant with a ≧25 and <50% decrease from baseline in total score.
Time Frame: From Baseline to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
Participants
  From baseline to Week 2: Responder | 2 | 4 | 2
  From baseline to Week 2: Partial responder | 9 | 3 | 4
  From baseline to Week 2: No response | 10 | 12 | 14
  From baseline to Week 4: Responder | 6 | 6 | 4
  From baseline to Week 4: Partial responder | 8 | 5 | 8
  From baseline to Week 4: No response | 7 | 8 | 8
  From baseline to Week 6: Responder | 11 | 6 | 7
  From baseline to Week 6: Partial responder | 3 | 8 | 4
  From baseline to Week 6: No response | 7 | 5 | 9
  From baseline to Week 7: Responder | 11 | 4 | 6
  From baseline to Week 7: Partial responder | 4 | 9 | 7
  From baseline to Week 7: No response | 6 | 6 | 7

8. Secondary Outcome: Number of Subjects With Suicidal Ideations Collected by Columbia-Suicide Severity Rating Scale (C-SSRS) From Baseline to Week 2, 4, 6 and 7 for Part II.
Description: The FDA has adopted the 11 categories defined in the C-SSRS (Category 1 to 5 for suicidal ideation , Category 6 to 10 for suicidal behavior, and Category 11 for self-injurious behavior without suicidal intent) as their standard.
  Number of subjects with Suicidal Ideation: The maximum suicidal ideation category (1-5 on the C-SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Time Frame: From screen to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
Participants
  Week 0 (baseline) | 1 | 1 | 4
  Week 2 | 2 | 1 | 4
  Week 4 | 0 | 1 | 3
  Week 6 | 1 | 1 | 3
  Week 7 | 2 | 2 | 4

9. Secondary Outcome: Number of Subjects With Suicidal Behaviors Collected by Columbia-Suicide Severity Rating Scale (C-SSRS) From Baseline to Week 2, 4, 6 and 7 for Part II.
Description: The FDA has adopted the 11 categories defined in the C-SSRS (Category 1 to 5 for suicidal ideation , Category 6 to 10 for suicidal behavior, and Category 11 for self-injurious behavior without suicidal intent) as their standard.
  Number of subjects with Suicidal Behavior: The maximum suicidal ideation category (6-10 on the C-SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
Time Frame: From screen to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
Participants
  Week 0 (baseline) | 0 | 0 | 0
  Week 2 | 0 | 0 | 0
  Week 4 | 0 | 0 | 0
  Week 6 | 0 | 0 | 0
  Week 7 | 0 | 0 | 0

10. Secondary Outcome: Clinical Global Impression Scale -Improvement (CGI-I) From Baseline to Week 2, 4, 6 and 7 for Part II.
Description: CGI-Improvement (CGI-I) is a 7-point scale which rates illness has improved or worsened relative to a baseline state from 1 (Very much improved) to 7 (Very much worse).
Time Frame: From Baseline to Week 2, 4, 6 and 7
Population: ITT population This Outcome Measure was conducted for Part II only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
Number analyzed (Participants) | 21 | 19 | 20
score on a scale
  From baseline to Week 2 | 3.0 (0.84) | 3.1 (1.03) | 3.4 (0.60)
  From baseline to Week 4 | 2.8 (0.94) | 3.1 (1.49) | 2.9 (0.85)
  From baseline to Week 6 | 2.8 (1.44) | 2.8 (1.18) | 2.9 (1.17)
  From baseline to Week 7 | 2.6 (1.03) | 2.9 (1.15) | 3.0 (1.03)

ADVERSE EVENTS:
Time Frame: Part I: 5 weeks Part II: 7 weeks
Arm/Group | Part I: 1 PDC-1421 Capsule | Part I: 2 PDC-1421 Capsule | Part II: 2 PDC-1421 Capsule | Part II: 1 PDC-1421 Capsule Plus 1 Placebo | Part II: 2 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/21 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/21 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 11/21 | 12/19 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I: 1 PDC-1421 Capsule (N=6) | Part I: 2 PDC-1421 Capsule (N=6) | Part II: 2 PDC-1421 Capsule (N=21) | Part II: 1 PDC-1421 Capsule Plus 1 Placebo (N=19) | Part II: 2 Placebo (N=20)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respirator tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parlpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT02395978/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02395978/SAP_000.pdf